CLINICAL TRIAL: NCT05906654
Title: Oregon Healthy Brain Research Network Collaborative Center (OrHBRN): Sharing History Through Active Reminiscence and Photo-imagery (SHARP) Pilot Program
Brief Title: Sharing History Through Active Reminiscence and Photo-imagery (SHARP) Pilot Program
Acronym: SHARP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Prevention
Other Study IDs: 00011936
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Change

STUDY DESIGN:
Intervention Model Description: 21 individuals without cognitive impairment engage in the study intervention over 24 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants engage in walking and conversational reminiscence three times per week
  Interventions: Behavioral: Sharing History through Active Reminiscence and Photo-imagery (SHARP)

INTERVENTIONS:
Behavioral: Sharing History through Active Reminiscence and Photo-imagery (SHARP) — Behavioral intervention to increase physical and social activity. In triads, participants walk 1-mile neighborhood routes three times per week and engage in image-based conversational reminiscence.
  Other Names: SHARP

SUMMARY:
SHARP is a neighborhood-based and technology-supported approach to brain health for older Black adults that integrates walking and image-prompted social reminiscence to maintain or improve brain health.

DETAILED DESCRIPTION:
The SHARP study tests the feasibility, usability, and cultural relevance of an android application-supported walking study for brain health among older Black adults. The SHARP walking application enables the seamless integration of the brain-healthy behaviors of walking, social engagement, and reminiscence. Methods: Over the course of 24 weeks in the rapidly gentrifying historically Black neighborhoods of Portland, Oregon, triads aim to complete three 1-mile walks per week. The SHARP application is preprogrammed with 72 themed, 1-mile routes, accessible via a group tablet device. At three points along each route, GPS-triggered "Memory Markers" (historical images of local Black culture) appear on the walking application, serving as prompts for conversational reminiscence as triads walk. Walking reminiscence sessions are recorded for inclusion into a digital oral history archive.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified African American
* > 55 years old
* A long-time resident (>10 cumulative years) of Portland's historically black neighborhoods (currently or in within the last 10 years)
* Without symptoms of and without a diagnosis of Alzheimer's Disease (they must be preclinical subjects),
* Without serious cognitive impairment and must score > 24 on the age-education adjusted Mini-Mental State Exam
* Has internet access in the home.
* Able to ambulate independently, without walking aids
* Able to sustain walking at a moderate pace for 45 minutes.

Exclusion Criteria

* Serious or unstable medical condition (such as, but not limited to, cardiovascular disease, pulmonary disease, or severe arthritis) where participation in the trial would, in the opinion of the investigator, pose a significant health risk to the subject.
* Diagnosis of Alzheimer's disease, vascular dementia, Parkinson's disease, or other dementing illness.

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Feasibility | 24 weeks
  Program readiness scale - how close is the program to being ready to deploy to other older Black Americans?

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carder, P., Croff, R., Tuttle, A., Towns, J. (2022) Walking and Talking: Recommendations for Doing Mobile Interviews with Older Adults. Journal of Aging and Environment, DOI: 10.1080/26892618.2022.2030844
- [Result] Croff RL, Witter Iv P, Walker ML, Francois E, Quinn C, Riley TC, Sharma NF, Kaye JA. Things Are Changing so Fast: Integrative Technology for Preserving Cognitive Health and Community History. Gerontologist. 2019 Jan 9;59(1):147-157. doi: 10.1093/geront/gny069. PMID 29961887
- [Derived] Croff R, Aron S, Wachana A, Fuller P, Mattek N, Towns J, Kaye J. Walking and Social Reminiscence in Gentrifying Neighborhoods: Feasibility and Impact on Cognitive, Physical, and Mental Health Among Older Black Adults in the SHARP Study. Gerontologist. 2024 Sep 1;64(9):gnae019. doi: 10.1093/geront/gnae019. PMID 38412543